CCF IRB #: 16-1643 Approval Date: 2/10/2019

Expiration Date: 2/9/2020

Version # 6

Date Submitted: May 29, 2018

# The Cleveland Clinic Foundation Consent to Participate in a Research Study

Study Title: Registry Based, Randomized Controlled Trial comparing Long-Term Results of Heavyweight versus Medium Weight Mesh in Ventral Hernia Repair

Principal Investigator: Michael J. Rosen, MD (216) 445-3441

You are being invited to participate in a research study. A research study is designed to answer specific questions about new ways to prevent, detect, and treat disease. Being in a research study is different from being a patient. The purpose of this document is to provide a written summary of the discussion and exchange of research information you had with the research team. It is also for use as a reference during the study.

#### Please note:

- You are being asked to participate in a research study
- Ask as many questions as needed so you can make an informed decision.
- Carefully consider the risks, benefits, and alternatives of the research
- Your decision to participate is completely voluntary and will have no effect on the quality of your medical care if you choose not to participate. You can also withdraw from the study at anytime.

## 1. INFORMATION ON THE RESEARCH

## Why are you being asked to take part in this research?

You are being asked to participate in a clinical research study because you are scheduled to undergo repair of your ventral hernia as part of your needed medical care.

## Why is the research study being done?

Your ventral hernia requires the use of mesh for repair. Currently, there are several different types of mesh available for use during ventral hernia repair. Synthetic mesh, which will be used for your ventral hernia repair, is divided into three categories based on its weight: light, medium, and heavy. The most common types of synthetic mesh used are mediumweight and heavyweight. There are proposed advantages and disadvantages to both mesh types, although these have not been proven. Specifically, heavyweight mesh is thought to be associated with increased postoperative pain and "stiff abdomen" while mediumweight mesh is thought to have a higher rate of ventral hernia recurrence. There is currently no consensus as to which mesh type is better, which is why we are doing this study.

## How many people will take part in this study?

Approximately 352 patients will be enrolled in this study at four institutions throughout the United States. We anticipate that approximately 200 patients will be enrolled in this study at the Cleveland Clinic Comprehensive Hernia Center. Patients enrolled in this study will be

Version # 6

Date Submitted: May 29, 2018

randomized to receive either heavyweight or mediumweight mesh at the time of their ventral hernia repair.

## What is involved if you decide to take part in this research study?

If you agree to be in this study, you will be asked to sign this consent form.

If you choose to take part in this study, we will review your medical records and ask you to fill out several short questionnaires that reflect your postoperative recovery during your postoperative clinic visits. These questionnaires should not take more than 15 minutes for you to fill out.

Your active participation in this study will last for 12 months and will involve one preoperative evaluation visit, one operative procedure visit, and 2 follow up visits.

If you agree to participate by signing the informed consent, you will have screening assessments completed. At this study visit, the doctor will ask about your past medical and surgical history and any medications you are taking and you will have a brief physical examination. If you qualify for study participation, you will be asked to join the study. If you choose to participate in the study, the study staff will collect additional information such as your gender, age, height, weight, your medical and surgical history, and information relating to your current ventral hernia. You will be asked to fill out baseline questionnaires at this appointment. The questionnaires will take approximately 15 minutes to complete.

You will receive routine preoperative care, which will be personalized for each patient. This routine care is not part of the study.

### Randomization

If you participate in this study, you will be assigned to a study group by chance using a process similar to the flip of a coin. This process is called randomization. This means that half of the people in this study will have their ventral hernia repaired with heavyweight synthetic mesh and half of the people in this study will have their ventral hernia repaired with mediumweight synthetic mesh. You will not know with which type of mesh your hernia will be repaired until the completion of your participation in this study. However, this information can be obtained if you have a medical emergency. Randomization will occur at the time of surgery. More precisely, randomization will occur at the moment your surgeon will place the mesh for your hernia repair. At this moment you will be assigned to receive either heavyweight or medium weight synthetic mesh.

### **Preoperative Visit**

This will be your first meeting with your surgeon. During this visit, your surgeon will evaluate you for a ventral hernia and determine if you are a surgical candidate for ventral hernia repair. If your surgeon believes that you are a candidate for ventral hernia repair and that you meet the criteria for this study, he/she will discuss this will you. You will be given this informed consent document and any questions that you have related to this study will be answered. Basic information about your health will be collected and physical examination will be performed.

Version # 6

Date Submitted: May 29, 2018

These are consistent with standard of care. As part of this study, you will be asked to fill out two questionnaires related to your quality of life and current pain.

### **Day of Surgery**

Your surgery will be performed in the usual manner, independent of your participation or not in this study. During the operation, you will be randomized to receive either heavyweight or medium weight synthetic mesh. As part of the study your doctor will collect information about your hernia or your surgery, such as the size of the ventral hernia, how long the surgery took, how much blood you lost during the surgery, antibiotics and IV fluids that are given, and how the ventral hernia was repaired. While this information is standard of care, it will also be used for study purposed.

## Follow-Up

You will be given instructions to return to the physician's clinic to be examined by the study doctor at one month and 12 months following your surgery. This time period for follow-up is standard of care. You will have your incisions and wounds evaluated and examined for general health and hernia recurrence. You will be asked about any medications you are taking and about any problems you may have had with your ventral hernia repair. Information about any admissions to the hospital or any subsequent procedures that may have been performed during this time will be collected. In addition to standard of care procedures, you will be asked to complete the same surveys that you filled out prior to surgery at each of these visits. You will be informed how your ventral hernia was repaired at the time of your 12 month follow-up appointment.

If at any time throughout the study period a ventral hernia recurrence is suspected clinically, then an abdominal CT scan will be performed to objectively evaluate the repair as standard of care dictates. All additional procedures, interventions, and adverse events will be collected throughout the final visit at 12 months postoperatively. The entire length of your active participation in this study will be for approximately 12 months following your hernia is repaired. In case you are not able to attend personally to your follow-up visit due to any reason, you have the option to follow-up with your surgeon using the Cleveland Clinic platform for Virtual Visits. The information from follow-up visits originated from this modality will also be used for this study. In case you are not able to have your visit with the surgeon 12 months after the surgery due to any reason, we will contact you over the telephone where you will be able to answer the same surveys.

### How long will you be in the study?

Your participation in this study will last for 12 months from the date of your original ventral hernia repair surgery. You can choose to stop participating at any time without penalty or loss of routine perioperative surgical care to which you are entitled. However, if you decide to stop participating in the study, it is important you talk with your doctor first.

#### 2. ALTERNATIVES

Version # 6

Date Submitted: May 29, 2018

## What are the alternatives to participation in the research study?

You do not have to take part in this study if you do not want to participate or your feel uncomfortable with any part of the aforementioned process. Your choice to participate or not will have no impact on the clinical care you will receive from your doctor. Should you decide to take part and later change your mind, you can do so at any time. Again, withdrawing from this research study will have no impact on the clinical care you will receive from your doctor.

#### 3. RISKS

## What are the risks of participating in the research study?

Questionnaires: It is possible that some of the questions may be upsetting or you may feel uncomfortable answering them. If you do not wish to answer a question or participate in a portion of the non-invasive testing, we will skip that portion of the study.

Personal Health Information: There is a small risk to the confidentiality of your data. Safeguards are in place to protect your information. Data will be stored on a password-protected computer at Cleveland Clinic that is accessible only to the study staff.

#### 4. BENEFITS

## What are possible benefits of participating in the research?

If you agree to take part in this study, there is NO direct medical benefit to you. We hope the information learned from this study will benefit medical science and provide information which may help improve the field of ventral hernia surgery.

## 5. COSTS

There will be no additional costs to you as a result of taking part in this study. However, routine medical care for your condition (the care you would receive whether or not you were in this study) will be charged to you and/or your insurance company. You will be responsible for any co-payments and deductibles that are standard for your insurance coverage.

## 6. COMPENSATION

### Are there any payments to you if you participate in this study?

There are no payments to you should you decide to participate in this study as all care is routine and standard of care for patients with a ventral hernia.

## 7. RESEARCH RELATED INJURY

### What will happen if you are injured as a result of taking part in the research?

In the event that you are injured as a result of participation in this research, medical care is available to you. The costs of such medical care will be billed to you or your insurance company. There are no plans to provide compensation for lost wages, direct, or indirect losses. The Cleveland Clinic will not voluntarily provide compensation for research related injury. You are

Version # 6

Date Submitted: May 29, 2018

not waiving any legal rights by signing this form. Further information about research related injury is available by contacting the Institutional Review Board at (216) 444-2924.

## 8. PRIVACY AND CONFIDENTIALITY

## What will happen to your information that is collected for this research?

Cleveland Clinic has rules and procedures to protect information about you. Federal and State Laws also protect your privacy.

The research team working on the study will collect information about you. This includes your health information, data collected for this research study, and personal identifying information including your name, address, date of birth, and other identifying information. This information will be used for the stated purpose of the study.

Generally, only people on the research team will know your identity and that you are in the research study. However, sometimes other people at Cleveland Clinic may see or give out your information. These included people who review research studies including the Institutional Review Board and Research Compliance, their staff, lawyers, or other Cleveland Clinic staff. If you agree, your personal physician may be informed of your participation in the study.

People outside of Cleveland Clinic may need to see your information for this study. Examples include government groups (such as the Food and Drug Administration) and safety monitors. Cleveland Clinic will do our best to ensure your information is kept confidential and that only the health information which is minimally required to conduct the study is used or disclosed to people outside Cleveland Clinic. However, people outside Cleveland Clinic who receive your information may not be covered by this promise.

You do not have to give this permission to use and give out your information. However, you will not be able to participate in this research study without providing this permission by signing this consent form. The use and disclosure of your information has no expiration date.

You may cancel your permission to use and disclose your information at any time by notifying the Principal Investigator in writing, Michael Rosen MD, 9500 Euclid Avenue, Cleveland, Ohio 44195. If you do cancel your permission to use and disclose your information, your participation in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in the study.

### 9. RESULTS

## What will happen to the results of this study?

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

If the results of this study are published, your identity will remain confidential.

Version # 6

Date Submitted: May 29, 2018

## 10. CONFLICT OF INTEREST

Do the researchers or institution have any conflicts of interest relating to this study? Yes, Dr. Rosen is the Founder and Chief Executive Officer of the Americas Hernia Society Quality Collaborative (AHSQC) Foundation. He receives a salary for these services. The AHSQC will receive and store data collected as part of this research project. These financial interests are being managed and are within permissible limits established by the Cleveland Clinic's Conflict of Interest Policy. If you have any questions regarding these conflicts of interests, please ask your doctor or call the Cleveland Clinic Institutional Review Board at (216) 444-2924.

## 11. QUESTIONS

## Who do you call if you have any questions or problems?

If you have any questions, concerns, or complaints about the research or develop a research-related problem, contact Michael J. Rosen, MD at (216) 445-3441 during regular business hours (8am-5pm). After hours, please call the clinic operator at (216) 444-2000 or (800) 223-2273 and ask for the General Surgery resident on call. If you have questions about your rights as a research subject, you may contact the local Cleveland Clinic Institutional Review Board at (216) 444-2924.

### 12. VOLUNTARY PARTICIPATION

# What are your rights as a research participant?

Taking part in this study is voluntary. You will be told of any new, relevant information from the research that may affect your health, welfare, or willingness to continue in this study. You may choose not to take part or may leave the study at any time. Withdrawing from the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to withdraw from the study you should discuss with your study doctor your decision to ensure a safe withdrawal.

You may refuse to be in or remove yourself from the study at any time without providing reason and this will not affect the standard of care you receive. To withdraw from the study, tell the principal investigator you no longer want to participate by contacting Michael Rosen, MD at 216-445-3441.

If you choose to withdraw from the study, you will be followed based on standard of care at your institution. The investigator can remove you from the study without your approval. Possible reasons could be if participation appears to be medically harmful to you, if it is discovered that you do not meet eligibility requirements, or if the study is cancelled.

Version # 6

Date Submitted: May 29, 2018

## 13. SIGNATURES

## Statement of participant

I have read and have had verbally explained to me the above information and have had all my questions answered to my satisfaction. I understand that my participation is voluntary and that I may stop my participation in the study at any time. Signing this form dose not waive any of my legal rights. I understand that a signed copy of this consent will be provided to me. By signing below, I agree to take part in this research study.

| Printed Name of Participant | | |
|---|---|---|
| Participant Signature | Date | |
| a discipant dignature | Butt | |
| Statement of person conducting informed I have discussed the information contained in opinion that the participant understands the with this research study. | n this document with the participant and it | - |
| Printed Name of Person Obtaining Consent | | |
| Simulation of Paragraph Obtaining Constant | Date | |
| Signature of Person Obtaining Consent | Date | |

| *1 |
|----|